CLINICAL TRIAL: NCT03458403
Title: Endoscopist and Endoscope Motions During Digestive Endoscopy
Acronym: EndoMouv
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IHU Strasbourg (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 17-001; 2017-A01968-45 (Other: ANSM France)
Record Dates: First submitted 2018-03-02; First posted 2018-03-08 (Actual); Last update posted 2023-02-28 (Actual); Status verified 2023-02

CONDITIONS: Scheduled Gastroscopy Under Sedation
Keywords: Digestive endoscopy; Tracking motion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Motions during gastroscopy (Experimental): Recording of endoscopist and endoscope motions right after the endoscopic exam the patient came for.
  Interventions: Procedure: Motions during gastroscopy

INTERVENTIONS:
Procedure: Motions during gastroscopy — Recording of endoscopist and endoscope motions right after the endoscopic exam the patient came for. The endoscope is removed halfway up the esophagus and inserted into the pylorus to the descending duodenum. The gesture is repeated three times.

SUMMARY:
The aim of the study is to record and analyze endoscopist and endoscope motions to identify key movements in flexible endoscopy.

DETAILED DESCRIPTION:
The increasing development of interventional digestive endoscopy raises the challenge to teach and learn complex endoscopic procedures. Nowadays experts are facing the challenge of explaining precisely an elaborate choreography of movements performed during the procedure, while novices are confronted with a broad range of hand, wrist and shoulder movements each resulting in different endoscope responses. The teaching strategy of endoscopy could benefit from a dedicated motion library that would associate the endoscopist's motion and the consequent endoscope response. A simplified endoscopic language made of individual motions could greatly shorten the learning curve.

The aim of the study is to record and analyze endoscopist and endoscope motions to identify key movements in flexible endoscopy.

ELIGIBILITY:
Inclusion Criteria:

* Patient over 18 years old
* Patient who are scheduled for a gastroscopy procedure under sedation
* Patient able to understand the study and provide written informed consent
* Patient affiliated to the French social security system.

Exclusion Criteria:

* Patient with an altered upper GI anatomy due to previous surgery
* Patient with a known anomaly of the upper GI anatomy
* Patient carrying an implantable medical device (pacemaker…)
* Patient with a condition preventing its participation to study procedures, according to investigator's judgment
* Pregnancy or breastfeeding
* Patient in custody
* Patient under guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2018-08-29 (Actual); Primary Completion 2022-01-28 (Actual); Study Completion 2022-01-28 (Actual)

PRIMARY OUTCOMES:
Body motions recording | At time of endoscopy
  Body motions recording using the Xsens tracking device. The Xsens motion tracking system consists of 17 wireless motion sensors that are applied with straps to the endoscopist without hindering natural movements.
Endoscope motions recording | At time of endoscopy
  Endoscope motions recording using the Aurora electromagnetic tracking system (NDI, Waterloo, Canada) inserted in the endoscope operating channel.
  The Aurora electromagnetic tracking system is designed for tracking tip and orientation of rigid and flexible endoscopes. The system consists of an electromagnetic field generator and a probe carrying the captors.
Endoscope wheels rotation recording | At time of endoscopy
  External video recording of the endoscope wheels rotation.
Endoluminal images recording | At time of endoscopy
  Endoluminal images recording using the endoscopic camera.

CONTACTS AND LOCATIONS:
Overall Officials: Silvana Perretta, MD, PhD, Principal Investigator — Service de Chirurgie Digestive et Endocrinienne - Nouvel Hôpital Civil - Strasbourg
Locations (1):
- Service de Chirurgie Digestive et Endocrinienne - Nouvel Hôpital Civil, Strasbourg, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kranzfelder M, Wilhelm D, Doundoulakis M, Schneider A, Bauer M, Reiser S, Meining A, Feussner H. A probe-based electromagnetic navigation system to integrate computed tomography during upper gastrointestinal endoscopy. Endoscopy. 2014 Apr;46(4):302-5. doi: 10.1055/s-0033-1358814. Epub 2013 Nov 19. PMID 24254384